CLINICAL TRIAL: NCT01671384
Title: Randomized Placebo Controlled Trial of Valproate and Levocarnitine in Children With Spinal Muscular Atrophy Aged 2-15 Years
Brief Title: Valproate and Levocarnitine in Children With Spinal Muscular Atrophy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Additional Professor, Department of Pediatrics, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Valproate and SMA
Record Dates: First submitted 2012-08-13; First posted 2012-08-23 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Spinal Muscular Atrophy
Keywords: Valproate; levocarnitine; SMA; physiotherapy; placebo
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Valproic Acid; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valproate, levocarnitine (Active Comparator): The patients will be randomized into two groups:
  Group I (Physiotherapy + Placebos) Group II (Physiotherapy + Valproate and Levocarnitine)
  Interventions: Drug: Valproate, Levocarnitine
- Placebo (Placebo Comparator): All patients will be randomized into two groups:
  Group I (Physiotherapy + Placebos) Group II (Physiotherapy + Valproate and Levocarnitine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valproate, Levocarnitine — All patients with diagnosis of SMA aged 2-15 years already registered in Myopathy Clinic of AIIMS will be recalled. Information will be sent to all Government Hospitals in Delhi that such a study is currently in progress and all the referrals will also be recruited. These patients and all those newly diagnosed at Myopathy Clinic, AIIMS will be randomized into two groups:
  Group I (Physiotherapy + Placebos) Group II (Physiotherapy + Valproate and Levocarnitine)
  The investigators will be blinded to the code of the medicine. It will be broken only at the end of the study or if there are any significant side effects. So one group will receive Valproate and levocarnitine and other group will receive Placebo and placebo.
  Other Names: Valprol and carnisure
  Arms: Valproate, levocarnitine
Drug: Placebo — All patients with diagnosis of SMA aged 2-15 years already registered in Myopathy Clinic of AIIMS will be recalled. Information will be sent to all Government Hospitals in Delhi that such a study is currently in progress and all the referrals will also be recruited. These patients and all those newly diagnosed at Myopathy Clinic, AIIMS will be randomized into two groups:
  Group I (Physiotherapy + Placebos) Group II (Physiotherapy + Valproate and Levocarnitine)
  The investigators will be blinded to the code of the medicine. It will be broken only at the end of the study or if there are any significant side effects. So one group will receive Valproate and levocarnitine and other group will receive Placebo and placebo.
  Other Names: Sugar based syrup
  Arms: Placebo

SUMMARY:
Spinal muscular atrophy (SMA), an autosomal recessive disorder, is characterized by muscle weakness due to degeneration of anterior horn cells in the spinal cord and brain stem nuclei. It has a variable incidence of 1 in 6700 to 1 in 25000 live births and prevalence of 0.12 to 25 per 10,000 populations in different geographic areas and genetic constitution. A homozygous deletion/mutation involving exon 7 in SMN1 (survival motor neuron 1) is present in around 95% of the cases, resulting in the biochemical deficiency of the SMN protein. A genomic duplication at the same locus produces nearly identical SMN2 (survival motor neuron 2) that differs from SMN1 by a nucleotide substitution that promotes exon 7 exclusion thus giving rise to only a fraction of the full length protein. Phenotypic variation in SMA correlates with the number of SMN2 gene copies and the level of SMN protein in cells.

Several hypotheses including defective inhibition of apoptosis, glutamate excitotoxicity and lack of a neurotrophic factor(s) in nerve or muscle have been speculated in the pathogenesis of SMA.

Valproic acid (VPA), a histone deacetylase (HDAC) inhibitor, directly increases SMN expression in SMA patient-derived cell lines in vitro. Till date 3 open label trials and 1 placebo controlled RCT of VPA in human subjects have been published, all indicating a possible benefit in strength and/or motor function. Till date there is no effective therapy for SMA. Therapy is mainly supportive and palliative which can prolong lifespan and prevent complications to some extent without actually curing the disease.

Children with SMA may have a reduced capacity to synthesis carnitine consequent to significantly diminished skeletal muscle mass. VPA independently inhibits carnitine transport and its metabolites deplete carnitine levels by binding to them. So along with valproate these patients should be supplemented with carnitine.

With this background the investigators have planned a double blind randomized placebo controlled trial of Valproate and levocarnitine in 60 children (30 each in intervention and control arm) with Spinal Muscular Atrophy aged 2-15 years over a 2 year period with one baseline and four follow up visits. The study will be conducted in the Department of Pediatrics, AIIMS at the Myopathy clinic.

DETAILED DESCRIPTION:
Spinal muscular atrophy is an autosomal recessive disease of varying severity that destroys motor neurons, resulting in atrophy and weakness of the voluntary muscles. Around 95% of the cases demonstrate a homozygous deletion/mutation involving exon 7 in SMN1 (survival motor neuron 1), resulting in the biochemical deficiency of the SMN protein.

Although the pathogenesis of the spinal muscular atrophy remains speculative, several hypotheses include defective inhibition of apoptosis, glutamate excitotoxicity and lack of a neurotrophic factor(s) in nerve or muscle.

Valproic acid (VPA), a histone deacetylase (HDAC) inhibitor, directly increases SMN expression in SMA patient-derived cell lines in vitro. It has also been demonstrated to have neuroprotective properties on glutamate induced excitotoxicity via up-regulation of alphasynuclein and increases neurite outgrowth in vitro.

The molecular genetic basis of spinal muscular atrophy (SMA), an autosomal recessive neuromuscular disorder, is the loss of function of the survival motor neuron gene (SMN1). The SMN2 gene, a nearly identical copy of SMN1, has been detected as a promising target for SMA therapy. Transcriptional SMN2 activation or modulation of its splicing pattern to increase FL-SMN levels is believed to be clinically beneficial and therefore a crucial challenge in SMA research. Drugs such as valproic acid, phenylbutyrate, and sodium butyrate that mainly act as histone deacetylase inhibitors can mediate both: they stimulate the SMN2 gene transcription and/or restore the splicing pattern, thereby elevating the levels of FL-SMN2 protein.

Till date 3 open label trials and 1 placebo controlled RCT of VPA in human subjects have been published, all indicating a possible benefit in strength and/or motor function.

Children with SMA may have a reduced capacity to synthesis carnitine consequent to significantly diminished skeletal muscle mass. VPA independently inhibits carnitine transport and its metabolites deplete carnitine levels by binding to them. So along with valproate these patients should be supplemented with carnitine.

Childhood spinal muscular atrophy (SMA) is a common autosomal recessive disorder, which is characterized by muscle weakness due to degeneration of motor neurons in the spinal cord and brain stem nuclei. Progression of the disease is due to loss of anterior horn cells, thought to be caused by apoptosis. Positional cloning strategies have revealed several gene candidates including the gene for the Survival Motor Neuron(SMN) and the neuronal apoptosis inhibitory protein (NAIP). Both genes are duplicated on chromosome 5.

The survival motor neuron transcript is encoded by two genes, SMNT and SMNC. The autosomal recessive proximal SMA that maps to 5q12 is caused by mutations in SMNT gene. SMNT exon 7 is not detected in approximately 95% of SMA cases because of either deletion or sequence conversion events.

Recently an international collaborative effort through the European Neuromuscular SMA Consortium, as noted above, has established diagnostic criteria.

1. Weakness is the central feature. The weakness should be symmetrical, proximal more than distal, and accompanied by hypotonia. The trunk is commonly involved. Weakness in the legs is characteristically greater than in the arms.
2. Denervation demonstrated by electromyography, muscle biopsy and clinical criteria. Recently, the presence of the survival motor gene defect has become accepted as a reliable diagnostic test for spinal muscular atrophy.

Possible therapeutic strategies include the use of motor neurotrophic agents, glutamate inhibitors, histone deacetylase inhibitors and embryonic grafts.

Valproate, a short chain fatty acid histone deacetylase inhibitor has been shown to increase the protein level of SMN2 by 2 to 4 fold through transcription activation and restoration of the correct splicing of SMN 2 via increased levels of Htra2-beta1 in fibroblast cell lines from SMA patients and it has also been shown to raise the SMN protein level also in neuronal tissue.11 Till date 3 open label trials and 1 placebo controlled RCT of VPA in human subjects have been published, all indicating a possible benefit in strength and motor function. Recently the results of CARNI-VAL (valproate and carnival) trial has been published. It is a multicentric trial with 2 parts. The 1st one is a double blinded placebo controlled randomised trial of 61 SMA patients aged 2 to 8 years. It has indicated possible benefit in motor function and strength in younger patients with favourable and normal BMI profile. The 2nd one is a prospective single armed trial of valproate and carnitine in 33 ambulatory children in SMA aged 3-17 years. No significant improvement was noted in muscle strength and functional status over 12 months period.

Valproate is an FDA approved drug used for more than three decades in epilepsy treatment. Common side effects are dyspepsia and / or weight gain. Less common side effects are dysphoria, fatigue, dizziness, drowsiness, hair loss, headaches, nausea, sedation and tremors. It also causes hyperammonemia. It has also been reported to cause blood dyscrasias, impaired liver function, jaundice, thrombocytopenia and prolonged coagulation times.

Because there has been no effective therapy for SMA, management till date consists of preventing or treating the complications. Complications of severe weakness include restrictive lung disease, poor nutrition, orthopedic deformities, immobility and psychosocial problems. Gene-specific therapy is not yet available. Noninvasive ventilation and percutaneous gastrostomy reportedly improves the quality of life with no effect on survival. The goal of active but nonfatiguing exercises is to maintain range of motion, increase muscle flexibility, and prevent contractures. Genetic counseling should be offered to all families of patient's with SMA.

Sample size This has been calculated with MMT as the primary outcome using repeated measures design (1 pre and 4 post measurements). Assuming mean ± SD MMT score in the control group at enrollment as 120± 55 (based on the baseline status of patients attending our routine myopathy clinic) and expecting an improvement of at least 30% in the intervention arm (i.e., 156± 55), with correlation coefficient as 0.6, 90% power and 5% 2 sided α (i.e., 95% CI), the investigators require a minimum of 25 cases in each group. Considering about 20% loss to follow up the investigators would enroll 30 children in each of the 2 study arms, i.e., a total of 60 cases.

Randomization: Block randomization with variable block size will be used to generate random numbers for allocation of study children in one of the two groups.

Interim analysis It will be done after 20 patients have been enrolled to assess efficacy of the drug. If efficacy is clear cut further continuation of the study will not be justified.

Patient recruitment

All patients with diagnosis of SMA aged 2-15 years already registered in Myopathy Clinic of AIIMS will be recalled. Information will be sent to all Government Hospitals in Delhi that such a study is currently in progress and all the referrals will also be recruited. These patients and all those newly diagnosed at Myopathy Clinic, AIIMS will be randomized into two groups:

Group I (Physiotherapy + Placebos) Group II (Physiotherapy + Valproate and Levocarnitine) Patients weighing less than 20 kg will receive liquid formulation of either sodium Valproateor placebo. Patients weighing more than 20 kg will receive oral tablets of either sodium Valproate/ placebo.

Day 1-Day 10 Day 11- Day 20 Day 21 onwards < 10 Kg 1 ml BD 2 ml BD 2 ml TDS 11-15 Kg 1.5 ml BD 2 ml TDS 3 ml TDS 16-20 Kg 2 ml BD 3 ml TDS 4 ml TDS 21-25 Kg 100 mg (1 tab BD) 200 mg (1 tab BD) 200 mg (1 tab TDS) 26-30 Kg 100 mg (1 tab TDS) 200 mg (1 tab TDS) 200 mg (2 -1-1) 31-35 Kg 100 mg (1 tab TDS) 200 mg (1 tab TDS) 200 mg (2-1-2) All patients in the intervention arm will be supplemented with Carnitine 50mg per kg per day (maximum 1000mg) in 2 divided doses during the entire period of valproate therapy .The other group will receive placebo.

The investigators will be blinded to the code of the medicine. It will be broken only at the end of the study or if there are any significant side effects.

Valproate is already being used for patients with epilepsy and has no significant side effects. Till date, besides conservative management no other treatment for SMA is available. This trial is thus justified.

Periodic evaluation of the data will be done by a Data Safety Management Board (DSMB) which will be comprised by eminent experts.

Informed consent It will be taken on a duly made consent form before starting the study. The patient or his parent's will have the right to withdraw from the study at any point of time with no disadvantage to the patient. No harmful effect is expected but in case of any research related injury, the best possible care at AIIMS will be provided.

A detailed history and physical examination will be carried out on a predesigned proforma. All children will undergo DNA testing for exon7 deletion of SMNT gene. All will have CPK levels and routine hemogram and liver function tests. If the exon7 deletion is absent, EMG, NCV and muscle biopsy will be performed. Baseline assessment will include a detailed muscle charting on a 5 point scale as per the principles of manual muscle testing by a child physiotherapist. Other tests will include functional measure using modified Hammersmith Functional Motor Scale (MHFMS) and forced vital capacity (FVC) wherever possible.

Patients will be clinically evaluated at 12, 24, 36 and 52 weeks by history, examination and a careful muscle charting. Other tests will include functional measure using modified Hammersmith Functional Motor Scale (MHFMS) and forced vital capacity (FVC) wherever possible. Compliance will be ensured at every visit by checking their medicine packets for leftover medicines. At 24 weeks and 52 weeks follow up routine hemogram, liver function tests and additionally at 52 weeks serum valproate levels will also be done.

MMT (manual muscle testing) score will be expressed as total score out of 340. Similarly modified Hammersmith Functional Motor Scale (MHFMS) score will be expressed as total score out of. FVC (Forced vital capacity) will be expressed in Litres. Serum Valproate levels will be expressed in mg/ml. Side effect profile of valproate will be expressed as incidence of patients with the symptoms mentioned above. Incidence of patients with low platelet count (less than 1.5lacs/mm3) and elevated liver enzymes (OT and PT more than 40U/ L) will be recorded. Mean± 2SD change in MMT score, MHFMS score and FVC at each visit will be analysed using Wilcockson ranksum test and T test.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-15 years having motor weakness, hypotonia and hyporeflexia with onset noticed after 6 months of age.
* Presence of exon7 deletion of SMNT gene. OR Normal/ mildly elevated CPK with electrodiagnostic characteristics suggestive of neurogenic weakness, normal motor and sensory nerve conduction velocities and muscle biopsy showing neurogenic atrophy and /or evidence of reinnervation.

Exclusion Criteria:

1. SMA type I, onset before 6 months of age.
2. Severely ill and unstable patients requiring life support system.
3. Other causes like cerebral palsy, Down syndrome, connective tissue disorders, metabolic disorders.
4. Pre-existing liver damage, bone marrow depression and coagulation disorders.
5. Use of medications or supplements which interfere with valproic acid and carnitine metabolism within 3 months of study enrollment.
6. Current use of either valproate or levocarnitine. If study subject is taking valproate and carnitine then patient must go through a washout period of 12 weeks before enrollment into the study

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in muscle power on a 5 point scale as per the principles of manual muscle testing at 12, 24, 36 and 52 weeks | Over 52 weeks with assessment at baseline, 12, 24, 36 and 52 weeks
  Baseline assessment will include a detailed muscle charting on a 5 point scale as per the principles of manual muscle testing by a child physiotherapist.Patients will be clinically re-evaluated at 12, 24, 36 and 52 weeks by a detailed muscle charting on a 5 point scale as per the principles of manual muscle testing by a child physiotherapist.

SECONDARY OUTCOMES:
a) Change in functional measure using modified Hammersmith Functional Motor Scale (MHFMS) score at 12, 24, 36 and 52 weeks 12, 24, 36 and 52 weeks. | Over 52 weeks starting from baseline folloowed by assessment at 12, 24,36 and 52 weeks
  Baseline functional status will be assessed using modified Hammersmith Functional Motor Scale (MHFMS) score. Change in functional measure using modified Hammersmith Functional Motor Scale (MHFMS) score will be measured at 12, 24, 36 and 52 weeks

OTHER OUTCOMES:
Change in Forced vital capacity (FVC) at 12, 24, 36 and 52 weeks. | Over 52 weeks with baseline assessment followed by re evaluation at 12, 24, 36 and 52 weeks
  Baseline Forced vital capacity (FVC) followed by change in Forced vital capacity (FVC) at 12, 24, 36 and 52 weeks will be measured.
Prevalence of various side effects of valproate (as mentioned below)in the subjects at 12, 24, 36 and 52 weeks. | At baseline followed by assessments at 12, 24, 36 and 52 weeks (as and when required)
  All patients will be assessed for side effect profile of valproate (dyspepsia, weight gain, dysphoria, fatigue, dizziness, drowsiness, hair loss, headaches, nausea, sedation and tremors) at 12, 24, 36 and 52 weeks.
Prevalence of abnormalities of Hemogram and Liver Function tests in the subjects at 24 and 52 weeks | At 24 weeks and at 52 weeks
  Hemogram and Liver Function tests of all recruited patients will be done at 24 and 52 weeks
Serum Valproate levels at 52 weeks | At 52 weeks completed
  Serum Valproate levels of all subjects will be done at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gulati Sheffali, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India